CLINICAL TRIAL: NCT02459444
Title: Safety and Efficacy of Inspiratory Muscle Training for Preventing Adverse Outcomes in Patients at Risk of Prolonged Hospitalization
Brief Title: Inspiratory Muscle Training and Hospital Complications
Acronym: IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Mansueto Gomes Neto, Physiotherapy course coordinator, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1163-0679
Record Dates: First submitted 2015-05-19; First posted 2015-06-02 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Muscle Weakness
Keywords: Respiratory Muscles; Muscle Weakness; Hospitalization; Length of Stay; Mortality
MeSH Terms: conditions — Muscle Weakness | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMT group and physiotherapy (Experimental): Inspiratory muscle training with POWERBREATHE an approximate load of 50 % of MIP , for 1 set of 30 breaths twice a day, 7 days a week for 4 weeks ( total 56 sessions). Associated with physiotherapy program.
  Interventions: Device: Powerbreathe; Other: Physiotherapy
- Sham IMT group (Placebo Comparator): Inspiratory muscle training with the same device in the experimental group , however without charge , for 1 set of 30 breaths twice a day, 7 days a week for 4 weeks ( total 56 sessions). Associated with physiotherapy program.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Device: Powerbreathe — Respiratory equipment for physiotherapy, offering to load muscles inspiratory
  Other Names: MODEL: CLASSIC LIGHT RESISTANCE; ANVISA: CLASS I 81001390001; MANUFACTURER: HAB INTERNATIONAL LTD - UNITED KINGDOM
  Arms: IMT group and physiotherapy
Other: Physiotherapy — This was contemplated cinesioterapia unloaded, muscle stretching, coughing technique, sedestração and ambulation if the participant was fit.
  Other Names: Concurrent training

SUMMARY:
The inspiratory muscle training (IMT) is a feasible and safe strategy for patients and athletes, your goal is to recondition the respiratory muscles, providing optimization of lung capacity, either for high performance sport as to support metabolic wear caused by illness. It is generally agreed the positive impact of the application of a TMI Protocol on maximal inspiratory pressure (MIP), this benefit encourages individuals sick since weaning from mechanical ventilation (MV), to the optimization of physical performance in cardiac and / or pulmonary rehabilitation. The TMI is based on the principles: the burden imposed on the muscle; the specificity of training; the reversibility of the gain and muscle atrophy.

DETAILED DESCRIPTION:
This prospective double-blind (patient and evaluator) randomised controlled trial compared the efficacy of inspiratory muscle training and inspiratory muscle training. The study protocol for this trial was described elsewhere. This study was conducted in accordance with Consolidated Standards of Reporting Trials recommendations. The trial was performed at the Roberto Santos General Hospital in Salvador, Bahia, Brazil. This study was approved by the institutional hospital ethics committee (approval reference number 03/2014). Before enrolment, written informed consent was obtained from participants or their legal guardians.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the hospital ward;
* At least two of the following risk factors for prolonged hospitalization: two or more comorbidities; sepsis; liver, lung, or kidney diseases; neoplasia; mechanical ventilation; and use of vasopressor or dialysis therapy.

Exclusion Criteria:

* Patients with a cognitive disability that made them unable to perform the respiratory training;
* Uncontrolled cardiac arrhythmias;
* Circulatory shock;
* Acute ischemic heart disease;
* acute respiratory failure (characterised by a partial pressure of arterial oxygen < 60 mmHg or a partial pressure of arterial carbon dioxide > 50 mmHg);
* neuromuscular disease or myopathies;
* diaphragmatic paresis or paralysis were excluded from the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
hospital inpatient complications | Discharge from hospital
  Follow-up during hospitalization

SECONDARY OUTCOMES:
respiratory muscle strength | After 4 weeks follow
  Measured with manometer for 3 reps.

OTHER OUTCOMES:
peripheral strength | four weeks
  Medical Research Council score
Functional Independence Measure questionnaire | Discharge from hospital
  Identifies said functional capacity
Index of Barthel | Discharge from hospital
  Identifies said functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Balbino V Nepomuceno, MD, Study Director — Federal University of Bahia
Locations (1):
- Mansueto Gomes Neto, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Background] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429
- [Result] Griffiths LA, McConnell AK. The influence of inspiratory and expiratory muscle training upon rowing performance. Eur J Appl Physiol. 2007 Mar;99(5):457-66. doi: 10.1007/s00421-006-0367-6. Epub 2006 Dec 22. PMID 17186299
- [Result] Hogan MC, Welch HG. Effect of altered arterial O2 tensions on muscle metabolism in dog skeletal muscle during fatiguing work. Am J Physiol. 1986 Aug;251(2 Pt 1):C216-22. doi: 10.1152/ajpcell.1986.251.2.C216. PMID 3740252
- [Result] Martin AD, Smith BK, Davenport PD, Harman E, Gonzalez-Rothi RJ, Baz M, Layon AJ, Banner MJ, Caruso LJ, Deoghare H, Huang TT, Gabrielli A. Inspiratory muscle strength training improves weaning outcome in failure to wean patients: a randomized trial. Crit Care. 2011;15(2):R84. doi: 10.1186/cc10081. Epub 2011 Mar 7. PMID 21385346
- [Derived] Nepomuceno BRV Jr, Barreto MS, Almeida NC, Guerreiro CF, Xavier-Souza E, Neto MG. Safety and efficacy of inspiratory muscle training for preventing adverse outcomes in patients at risk of prolonged hospitalisation. Trials. 2017 Dec 28;18(1):626. doi: 10.1186/s13063-017-2372-y. PMID 29282152